CLINICAL TRIAL: NCT02959125
Title: NutFish and Nutrient Supplementation in Pregnancy Class to Improve Maternal and Birth Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Semarang Health Polytechnic (Other)
Responsible Party: Principal Investigator, Kun Aristiati Susiloretni, Dr, Semarang Health Polytechnic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SemarangHP
Record Dates: First submitted 2016-08-27; First posted 2016-11-08 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Pregnancy; Protein-Energy Malnutrition; Anemia
MeSH Terms: conditions — Protein-Energy Malnutrition; Anemia | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Intervention
  * NutFish based supplementation for 60 days
  * Multiple micro nutrient for 60 days
  * Health education in pregnancy class
  Interventions: Other: NutFish Based Food Supplementation; Dietary Supplement: Multiple micronutrients; Behavioral: Health Education in Pregnancy Class
- Control (Active Comparator): Control
  * Government food supplementation for 60 days
  * Iron Folic acid for 60 days
  * Health education in pregnancy class
  Interventions: Behavioral: Health Education in Pregnancy Class; Other: Government Food Supplementation; Dietary Supplement: Fe Supplementation

INTERVENTIONS:
Other: NutFish Based Food Supplementation — Cookies contain 500 Calories and 15 gram protein make from nut and ocean fish
  Arms: Intervention
Dietary Supplement: Multiple micronutrients — Vitamin A 5000 iu, vitamin D 400 iu, vitamin C 100 mg, vitamin B1 7.5 mg, vitamin B2 3 mg, vitamin B6 10 mg, vitamin B12 10 mcg, fluoride 1 mg, Fe fumarate 91 mg, niacinamide 20 mg, Ca pantothenate 7.5 mg, folic acid 400 mcg, Zn 5 mg, Ca lactate 250 mg, copper 0.1 mg, iodine 0.1 mg
  Arms: Intervention
Behavioral: Health Education in Pregnancy Class — Health education on pregnancy, complication, and breastfeeding by research team members
  Other Names: Intervention
Other: Government Food Supplementation — Cookies contain 500 Calories and 5 gram protein make from flour and egg
  Arms: Control
Dietary Supplement: Fe Supplementation — Ferrous Fumarate 60mg and folic acid 0.400 mg
  Arms: Control

SUMMARY:
This study evaluates the intervention of Nut Fish based food, micro nutrients supplementation and pregnancy class to improve maternal and birth outcome. This is cluster randomized trial with two arms. The intervention group will receive Nut Fish based supplementation, multiple micro nutrients, and pregnancy class. The control group will receive government food supplementation, iron folic acid supplementation, and pregnancy class.

DETAILED DESCRIPTION:
Objectives: To investigate whether a nut fish based food and dietary supplementation delivered to pregnant mothers with health education would benefit maternal and birth outcomes compared with the government standard of care.

Design. A randomized control trial will be implemented in rural community in Indonesia.

Intervention. The 2 trial arms will be control group (government standard of care) and intervention group with nut fish based food and dietary supplementation and health education series in the pregnancy class. A control group will receive government food supplementation package, Iron Folic acid pills and pregnancy class. An intervention group will receive NutFish based food supplementation, multiple micro nutrients, and pregnancy class. As a pilot study, all the intervention packages will be delivered by research team members.

Subjects. A total 72 first trimester of pregnant mothers will be enrolled with 36 pregnant mothers each group.

Outcome measures. Maternal outcome at 1 and 2 month after intervention namely weight increment, energy and protein intake, mid upper arm circumference, and complications. Birth outcomes include APGAR score, birth weight and length, preterm birth.

Analysis. Linear, logistic and multinomial logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* First trimester of pregnancy
* Anemic or Mid Upper Arm Circumference < 23.5cm or no weight gain
* Plan to deliver at village midwives
* residence in the study area

Exclusion Criteria:

* severe anemia < 7.0g/dl

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-10-30 (Estimated); Study Completion 2017-12-20 (Estimated)

PRIMARY OUTCOMES:
Birth weight | at delivery
  Infant weight (in grams) at birth

SECONDARY OUTCOMES:
APGAR score | at delivery
  Five criteria used as an index of health in the immediate neonatal period : Appearance, Pulse, Grimace, Activity, Respiration
Preterm birth | at delivery
  Delivery before 37 weeks gestation
Birth length | at delivery
  Infant length (in centimeters) at birth
Mid upper arm circumference | baseline, 30 (+/- 3), and 60 (+/- 3) days
  measured in centimeters, at the mid-point between the tip of the shoulder and the tip of the elbow
Gestational weight gain | baseline, 30 (+/- 3), and 60 (+/- 3) days
  Weight gained during pregnancy as compared to medical recommendation
Dietary intake | baseline, 30 (+/- 3), and 60 (+/- 3) days
  % nutrient intake compare to estimated average requirements (EAR). Dietary intake: energy, protein, zinc, Fe
Problems experience | baseline, 30 (+/- 3), and 60 (+/- 3) days
  Number of problems(minor and serious) experience by the mother during pregnancy. Minor problems include: backache, constipation, cramp, feeling faint, hot, headache, etc. Serious problem: Slow-growing babies, Vaginal bleeding, Deep vein thrombosis, High blood pressure, pre-eclampsia, etc We will aggregate in minor and serious problems

CONTACTS AND LOCATIONS:
Overall Officials: Kun A Susiloretni, Dr, Principal Investigator — Semarang Health Polytechnic
Locations (2):
- Indonesia (2):
  - Demak District Health Office, Demak, Central Java
  - Public Health Center of Karangawen 2, Demak, Central Java

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ota E, Hori H, Mori R, Tobe-Gai R, Farrar D. Antenatal dietary education and supplementation to increase energy and protein intake. Cochrane Database Syst Rev. 2015 Jun 2;2015(6):CD000032. doi: 10.1002/14651858.CD000032.pub3. PMID 26031211
- [Result] Imdad A, Bhutta ZA. Maternal nutrition and birth outcomes: effect of balanced protein-energy supplementation. Paediatr Perinat Epidemiol. 2012 Jul;26 Suppl 1:178-90. doi: 10.1111/j.1365-3016.2012.01308.x. PMID 22742610
- [Result] Haider BA, Bhutta ZA. Multiple-micronutrient supplementation for women during pregnancy. Cochrane Database Syst Rev. 2015 Nov 1;2015(11):CD004905. doi: 10.1002/14651858.CD004905.pub4. PMID 26522344